CLINICAL TRIAL: NCT06317142
Title: Investigating Disturbances in Glucose and Glycogen Dynamics in Prediabetes
Brief Title: Glucose and Glycogen Dynamics in Prediabetes
Acronym: GGD
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL84574.068.23
Record Dates: First submitted 2023-08-07; First posted 2024-03-19 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — acipimox

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy overweight volunteers: This group includes 15 healthy overweight volunteers. These participants will undergo two test days with one overnight stay. During these days several tests will be conducted including measurements such as muscle and liver glycogen, whole-body gluconeogenesis, substrate oxidation and postprandial hepatic and muscle glucose uptake will be assessed by 18F-FDG PET combined with an oral glucose tolerance test.
- Prediabetes volunteers-IFG: This group will include 15 subjects with impaired fasting glucose (IFG). These participants will undergo two test days with one overnight stay. During these days several tests will be conducted including measurements such as muscle and liver glycogen, whole-body gluconeogenesis, substrate oxidation and postprandial hepatic and muscle glucose uptake will be assessed by 18F-FDG PET combined with an oral glucose tolerance test.
  A subset of IFG prediabetes individuals with impaired fasting glucose (first 10 subjects enrolled) will receive a 4-day Acipimox treatment (3x 250mg capsules for three days (one with breakfast, one with lunch and one with snack) and 1x 250mg in the morning of day 4. After the intervention the participants will come to the university for two days with an overnight stay for tests (muscle and liver glycogen, whole-body gluconeogenesis, substrate oxidation, oral glucose tolerance test).
  Interventions: Drug: Acipimox 250 mg Oral Capsule
- Prediabetes volunteers-IGT: This group will include 15 subjects with impaired glucose tolerance (IGT). These participants will undergo two test days with one overnight stay. During these days several tests will be conducted including measurements such as muscle and liver glycogen, whole-body gluconeogenesis, substrate oxidation and postprandial hepatic and muscle glucose uptake will be assessed by 18F-FDG PET combined with an oral glucose tolerance test.
  A subset of IGT prediabetes individuals with impaired fasting glucose (first 10 subjects enrolled) will receive a 4-day Acipimox treatment (3x 250mg capsules for three days (one with breakfast, one with lunch and one with snack) and 1x 250mg in the morning of day 4. After the intervention the participants will come to the university for two days with an overnight stay for tests (muscle and liver glycogen, whole-body gluconeogenesis, substrate oxidation, oral glucose tolerance test).
  Interventions: Drug: Acipimox 250 mg Oral Capsule

INTERVENTIONS:
Drug: Acipimox 250 mg Oral Capsule — A subset of prediabetes individuals (first 10 IFG and 10 IGT subjects enrolled) will receive a 4-day Acipimox treatment (3x 250mg capsules for three days (one with breakfast,one with lunch and one with snack) and 1x 250mg in the morning of day 4.
  Other Names: Olbetam 250 mg oral capsule
  Groups: Prediabetes volunteers-IFG; Prediabetes volunteers-IGT

SUMMARY:
The goal of this observational study is to investigate changes in nocturnal and postprandial glucose and glycogen metabolism in individuals with impaired fasting glucose and impaired glucose tolerance compared to healthy, non-diabetic, overweight participants (15 per group). In addition, it will be investigated if reducing gluconeogenesis, by using the challenge agent Acipimox, in people with prediabetes can increase glucose tolerance and fat oxidation by increased reliance on hepatic glycogen. The main questions this project aims to answer are:

* whether there are differences in nocturnal glucose/glycogen metabolism in individuals with impaired fasting glucose, impaired glucose tolerance and healthy overweight controls.
* whether there are differences in postprandial glucose/glycogen metabolism in individuals with impaired fasting glucose, impaired glucose tolerance and healthy overweight controls.

Participants will visit the university for a screening visit and a visit with overnight stay for measurements of gluconeogenesis, glycogen, and substrate oxidation. A subgroup will receive [18F]-FDG to assess tissue-specific postprandial glucose uptake. Thereafter, 20 prediabetic individuals will follow a 4-day treatment with acipimox to decrease gluconeogenesis, followed by a second overnight visit with similar measurements as mentioned for the first visit.

ELIGIBILITY:
Inclusion Criteria for all groups:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Participants should have suitable veins for cannulation or repeated venipuncture
* Women are post-menopausal (defined as at least 1 year post cessation of menses)
* Aged ≥ 45 and ≤ 75 years
* Body mass index (BMI) 27 - 38 kg/m2
* Stable dietary habits (no weight loss or gain >5kg in the past 3 months)
* Sedentary lifestyle (not more than 2 hours of sports per week)

Inclusion Criteria for Prediabetic groups specifically:

Impaired Fasting Glucose: fasting blood glucose between 6.1 and 6.9 mmol/L and 2-h plasma glucose after ingestion of 75g oral glucose load below 7.8 mmol/L Impaired Glucose Tolerance: fasting blood glucose below 6.1 mmol/L and 2-h plasma glucose after ingestion of 75g oral glucose load between 7.8 and 11.1 mmol/L

Exclusion Criteria for all groups:

* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the Investigator
* Previously diagnosed with type 2 diabetes
* Patients with congestive heart failure and/or severe renal (eGFR <50mL/min) and or liver insufficiency or another condition that may interfere with outcomes measured in this study.
* Any contra-indication MRI scanning
* Alcohol consumption of >2 servings per day for men and >1 servings per day for woman
* Smoking in the past 6 months
* Medication use that may influence main outcome parameters, specifically the following types of medication: Type 2 diabetes medication, corticosteroids, thyroid medication.
* Participation in research or medical examination that included PET scanning in the last 3 months

Exclusion Criteria for Healthy overweight specifically:

- Any of the criteria mentioned above to define prediabetes

Exclusion Criteria for Prediabetic groups who will undergo acipimox treatment:

* Gout
* Hypersensitivity to acipimox or to any of the excipients in the tablet
* Peptic ulcer/dyspepsia
* Medication that interferes with Acipimox (statins, fibrates).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 healthy overweight participants, 15 participants with prediabetes characterised by IGT and 15 participants with prediabetes characterised by IFG. All participants will be aged 45-75y, with a BMI between 27-38 kg/m2, stable dietary habets, a sedentary lifestyle and no sign of active disease or excesive alcohol consumption.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Hepatic and muscle glycogen measured by 13Carbon-Magnetic resonance spectroscopy (13C-MRS) | During day 1 and day 2
  Difference in overnight and postprandial change of hepatic and muscle glycogen measured by 13C-MRS between healthy overweight volunteers and volunteers with IFG and IGT
Whole body gluconeogenesis determined by deuterated water | During day 1 and day 2
  Difference in whole-body gluconeogenesis between healthy overweight volunteers and IFG and IGT volunteers
Postprandial hepatic and muscle glucose uptake determined by Fluorodeoxyglucose-Positron emission tomography ([18F]-FDG-PET) combined with oral glucose tolerance test (OGTT) | During day 2
  Difference in glucose uptake between healthy overweight volunteers and IFG and IGT volunteers

SECONDARY OUTCOMES:
Oral glucose tolerance after acipimox treatment measured by OGTT | During day 2 and day 6
  Difference in glucose tolerance measured by OGTT before and after 4 days of acipimox treatment in prediabetic volunteers (intra- and inter-group comparisons)
Hepatic glycogen after acipimox treatment measured by 13C-MRS | During day 1,2, 5 and 6
  Difference in overnight change of hepatic glycogen before and after 4 days of acipimox treatment in prediabetic volunteers (intra- and inter-group comparisons)
Whole body gluconeogenesis after acipimox treatment determined by deuterated water | During day 1,2, 5 and 6
  Difference in whole body gluconeogenesis before and after 4 days of acipimox treatment in prediabetic volunteers (intra- and inter-group comparisons)

OTHER OUTCOMES:
Hepatic acetylcarnitine as a measure for hepatic gluconeogenesis determined by H-MRS | During day 1,2, 5 and 6
  Difference in hepatic acetylcarnitine between healthy overweight volunteers and individuals with IGT and IFG and the difference in hepatic acetylcarnitine before and after 4 days of acipimox treatment in prediabetic volunteers (intra- and inter-group comparisons).
Substrate oxidation (fat and carbohydrate oxidation) determined by indirect calorimetry | During day 1,2, 5 and 6
  Difference in substrate oxidation (fat and carbohydrate oxidation) between healthy overweight volunteers and IFG and IGT volunteers and the difference in substrate oxidation before and after 4 days of acipimox treatment in IFG and IGT volunteers (intra- and inter-group comparisons).
Dynamic water relaxation measurements with 1H-MRS (surrogate glycogen) | During day 1,2, 5 and 6
  Difference in water relaxation measures between healthy overweight volunteers and IFG and IGT volunteers.
Anthropometric measurements | During the screening day
  weight and height will be combined to report BMI in kg/m^2 (to characterize participants)
Body composition determined by Bodpod | During day 1
  fat mass and fat free mass as % (to characterize participants)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data can be obtained with the PI on request